CLINICAL TRIAL: NCT07309393
Title: Impact of Sugammadex Versus Neostigmine on Early Postoperative Pulmonary Function After Thoracoscopic Lung Resection: A Multicenter, Randomized, Double-Blind, Controlled Trial
Brief Title: Impact of Sugammadex Versus Neostigmine on Early Postoperative Pulmonary Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Shiyou Wei, Department of Anesthesiology, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025LY0107
Record Dates: First submitted 2025-08-03; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Residual Neuromuscular Block
Keywords: Sugammadex; Neostigmine; Forced Expiratory Volume (FEV1); Lung Resection; Quality of Recovery
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, controlled trial with parallel group assignment. Eligible patients undergoing unilateral thoracoscopic lung segmentectomy (not exceeding one lung segment) are randomized in a 1:1 ratio to receive either sugammadex (experimental group) or neostigmine plus atropine (control group) for reversal of rocuronium-induced neuromuscular blockade at the end of surgery. The primary focus is on comparing the effects on early postoperative pulmonary function recovery, with assessments conducted preoperatively and at postoperative 1 hour, 1-3 days, or before discharge.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind masking is implemented for participants and investigators to minimize bias. At the end of surgery, an independent anesthesia nurse prepares the study drug (sugammadex 2 mg/kg or neostigmine 0.03 mg/kg plus atropine 0.015 mg/kg) diluted in normal saline to a total volume of 10 mL in identical syringes, ensuring that the administering anesthesiologist and other study personnel remain blinded to the group assignment. Participants are also unaware of the assigned reversal agent. Blinding is maintained throughout the postoperative follow-up period, with unblinding reserved for emergencies or serious adverse events as per protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex Group (Experimental): Participants in this experimental arm receive sugammadex (2 mg/kg IV) for reversal of rocuronium-induced neuromuscular blockade at the end of unilateral thoracoscopic lung segmentectomy surgery. The drug is prepared by an independent anesthesia nurse, diluted in normal saline to 10 mL, and administered when the patient shows signs of awakening (e.g., TOF ratio 0.4-0.9 or full awakening). This arm includes 120 participants randomized in a 1:1 ratio. Postoperative assessments focus on pulmonary function recovery, pain, and complications.
  Interventions: Drug: Sugammadex
- Neostigmine Group (Active Comparator): Participants in this active comparator arm receive neostigmine (0.03 mg/kg IV) plus atropine (0.015 mg/kg IV) for reversal of rocuronium-induced neuromuscular blockade at the end of unilateral thoracoscopic lung segmentectomy surgery. The drugs are prepared by an independent anesthesia nurse, diluted in normal saline to 10 mL, and administered when the patient shows signs of awakening (e.g., TOF ratio 0.4-0.9 or full awakening). This arm includes 120 participants randomized in a 1:1 ratio. Postoperative assessments focus on pulmonary function recovery, pain, and complications.
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — Sugammadex is administered intravenously at a dose of 2 mg/kg for reversal of rocuronium-induced neuromuscular blockade at the end of unilateral thoracoscopic lung segmentectomy surgery. The drug is prepared by an independent anesthesia nurse, diluted in normal saline to a total volume of 10 mL in an identical syringe to maintain blinding. Administration occurs when the patient shows signs of awakening (e.g., TOF ratio 0.4-0.9 or full awakening). This is a single-dose intervention given once at the conclusion of surgery. Associated with the Sugammadex Group (experimental arm).
  Other Names: HengShu, Sugammadex sodium
  Arms: Sugammadex Group
Drug: Neostigmine — Neostigmine (0.03 mg/kg) combined with atropine (0.015 mg/kg) is administered intravenously for reversal of rocuronium-induced neuromuscular blockade at the end of unilateral thoracoscopic lung segmentectomy surgery. The drugs are prepared by an independent anesthesia nurse, diluted in normal saline to a total volume of 10 mL in an identical syringe to maintain blinding. Administration occurs when the patient shows signs of awakening (e.g., TOF ratio 0.4-0.9 or full awakening). This is a single-dose intervention given once at the conclusion of surgery. Associated with the Neostigmine Group (active comparator arm).
  Other Names: Neostigmine methylsulfate
  Arms: Neostigmine Group

SUMMARY:
Residual neuromuscular blockade (NMB) after general anesthesia increases the risk of postoperative respiratory complications (atelectasis, pneumonia, re-intubation) and delays pulmonary function recovery. Sugammadex, a γ-cyclodextrin that directly encapsulates rocuronium, reverses NMB rapidly and completely without cholinergic side effects, whereas neostigmine requires co-administration of an antimuscarinic and may leave residual blockade. In this multicenter, randomized, double-blind, controlled trial, 240 adult patients (ASA I-III) undergoing elective thoracoscopic lung resection (≤ 1 segment) will be randomized 1:1 to receive sugammadex (2 mg/kg) or neostigmine (0.03 mg/kg) + atropine (0.015 mg/kg) at the end of surgery. The primary endpoint is the percent decline in forced expiratory volume in 1 second (FEV₁) at 1 hour post-extubation compared to preoperative baseline; a ≥ 5% improvement with sugammadex is hypothesized. Secondary endpoints include FEV₁ at days 1-3, pain scores, opioid consumption, gastrointestinal recovery, quality of recovery (QoR-15), neuromuscular monitoring (TOF ratio), and incidence of postoperative pulmonary and surgical complications.

DETAILED DESCRIPTION:
Detailed Description:

Background: Thoracoscopic lung surgery requires general anesthesia with double-lumen endotracheal intubation and muscle relaxants to facilitate lung isolation and surgical exposure. Residual neuromuscular blockade after surgery can cause complications such as airway obstruction, atelectasis, pneumonia, prolonged PACU stay, and reduced patient satisfaction. Neostigmine, a commonly used acetylcholinesterase inhibitor, reverses neuromuscular blockade by increasing acetylcholine but may cause cholinergic side effects, requiring atropine co-administration. Sugammadex, a γ-cyclodextrin compound, encapsulates and inactivates rocuronium directly, reversing blockade without affecting cholinergic receptors and avoiding related adverse events. Sugammadex can also shorten operation time and improve turnover efficiency in thoracoscopic surgery.

Purpose: This study aims to compare the effects of sugammadex and neostigmine on early postoperative pulmonary function recovery in patients undergoing thoracoscopic lung resection, providing reliable clinical data to improve surgical management and enhance recovery.

Design: Patients planned for unilateral thoracoscopic lung segmentectomy will be randomized 1:1 to receive either sugammadex or neostigmine plus atropine for reversal of rocuronium-induced neuromuscular blockade at the end of surgery. Pulmonary function will be assessed using a portable spirometer before surgery and at postoperative 1 hour, 1 to 3 days, or before discharge. Other outcomes including postoperative pain, opioid consumption, gastrointestinal recovery, incidence of nausea/vomiting, quality of recovery (QoR-15 scale) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective unilateral thoracoscopic partial lung resection, with expected resection not exceeding one lung segment.
* Age between 18 and 80 years.
* American Society of Anesthesiologists (ASA) Physical Status classification I-III.

Exclusion Criteria:

* Contraindications to drug use, such as history of allergy, epilepsy, angina, ventricular tachycardia; contraindicated in patients with mechanical intestinal obstruction or urinary tract obstruction; contraindicated in cases of arrhythmia, bradycardia (<50 beats per minute), hypotension, or increased vagal tone; contraindicated in patients currently using depolarizing muscle relaxants (e.g., succinylcholine).
* Inability to correctly cooperate with portable lung function testing.
* Hepatic or renal insufficiency.
* Pregnancy, lactation, potential for pregnancy, or planning pregnancy.
* Preoperative history of drug abuse or addiction.
* Actual surgical resection exceeding one lung segment.
* Second surgery during postoperative hospitalization.
* Patients who refuse to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Forced Expiratory Volume in 1 Second (FEV1) from Baseline to 1 Hour Postoperatively | Preoperative (baseline, within 7 days before surgery) and 1 hour postoperative.
  The percentage decline in FEV1 (measured using a portable spirometer) at 1 hour after unilateral thoracoscopic lung segmentectomy surgery, compared to the preoperative baseline value. FEV1 represents the volume of air exhaled in the first second of a forced expiratory maneuver. The decline is calculated as [(preoperative FEV1 - postoperative FEV1) / preoperative FEV1] × 100%. A smaller decline indicates better early postoperative pulmonary function recovery.

SECONDARY OUTCOMES:
Change in Forced Expiratory Volume in 1 Second (FEV1) from Baseline to Later Postoperative Time Points | Preoperative (baseline, within 7 days before surgery) and postoperative day 1-3 or before discharge.
  The percentage decline in FEV1 (measured using a portable spirometer) at postoperative day 1-3 or before discharge, compared to the preoperative baseline value. FEV1 represents the volume of air exhaled in the first second of a forced expiratory maneuver. The decline is calculated as [(preoperative FEV1 - postoperative FEV1) / preoperative FEV1] × 100%. A smaller decline indicates better postoperative pulmonary function recovery.
Postoperative Pain Score | Postoperative 1 hour and postoperative day 1-3.
  Postoperative pain intensity assessed using the Verbal Response Scale (VRS), the score ranges from 0 to 10, with a total of 11 numbers corresponding to different pain levels: 0 indicates no pain; 1-3 indicates mild pain (tolerable and does not affect sleep); 4-6 indicates moderate pain (significant, affects sleep, and requires medication for relief); and 7-10 indicates severe pain (intense, intolerable, and severely affects life).

OTHER OUTCOMES:
Cumulative Opioid Consumption | Postoperative day 1-2 (up to 48 hours after surgery).
  Total cumulative opioid dosage (in morphine equivalents) administered postoperatively, including patient-controlled analgesia and rescue doses .
Neuromuscular Recovery (TOF Ratio) | At the end of surgery and 1 hour postoperative.
  Train-of-Four (TOF) ratio measured using a neuromuscular monitor on the ulnar nerve at the end of surgery. The TOF ratio is recorded as T4/T1, with a ratio ≥0.9 indicating complete neuromuscular recovery from rocuronium-induced blockade.
Gastrointestinal Function Recovery | Postoperative day 1-3.
  The time to first postoperative gastrointestinal flatus
Quality of Recovery (QoR-15 Score) | Postoperative day 1-3
  Postoperative recovery quality assessed using the Quality of Recovery-15 (QoR-15) questionnaire, a patient-reported scale covering emotional state, physical comfort, psychological support, physical independence, and pain. Scores range from 0 to 150, with higher scores indicating better recovery quality.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lv, PhD, Study Director — Shanghai Pulmonary Hospital, Tongji University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No